CLINICAL TRIAL: NCT07345507
Title: Comparison of Efficacy of Metformin Gel 30% vs Triple Combination Cream (Hydroquinone 4%, Flucinolone Acetonide 0.01%, Tretinoin 0.025%) in Treatment of Melasma in Tertiary Care Hospital Karachi.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Dr Summiya Shakeel Ahmed, FCPS part 2 Trainee dermatology, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: F.2-81/2024-GENL/24/JPMC
Record Dates: First submitted 2025-07-09; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Melasma
Keywords: Melasma; Efficacy; METFORMIN GEL; HYDROQUINONE 2%; TRETINOIN 0.025%
MeSH Terms: conditions — Melanosis | interventions — hydroquinone; Tretinoin

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (TRIPLE COMBINATION THERAPY GROUP) (Active Comparator): Triple combination cream (hydroquinone 2% + tretinoin 0.025% + fluocinolone acetonide 0.01%) applied nightly for 12 weeks. All participants also used broad-spectrum sunscreen (SPF ≥30) during daytime.
  Interventions: Drug: Triple combination cream (hydroquinone 2% + tretinoin 0.025% + fluocinolone acetonide 0.01%); Drug: Broad-spectrum sunscreen (SPF ≥30)
- Group B ( METFORMIN 30% GEL THERAPY GROUP ) (Experimental): Participants will apply 30% metformin gel topically to melasma-affected areas once nightly for 12 weeks. All participants will also use broad-spectrum sunscreen (SPF ≥30) during daytime.
  Interventions: Drug: Metformin gel, 30%; Drug: Broad-spectrum sunscreen (SPF ≥30)

INTERVENTIONS:
Drug: Metformin gel, 30% — Participants will apply 30% metformin gel topically to melasma-affected areas once nightly for 12 weeks. All participants will also use broad-spectrum sunscreen (SPF ≥30) during daytime.
  Arms: Group B ( METFORMIN 30% GEL THERAPY GROUP )
Drug: Triple combination cream (hydroquinone 2% + tretinoin 0.025% + fluocinolone acetonide 0.01%) — Topical triple combination cream containing hydroquinone 2%, tretinoin 0.025%, and fluocinolone acetonide 0.01%, applied once nightly to affected facial areas for 12 weeks
  Arms: Group A (TRIPLE COMBINATION THERAPY GROUP)
Drug: Broad-spectrum sunscreen (SPF ≥30) — Applied during daytime throughout the 12-week treatment period (both arms)

SUMMARY:
This study will compare two topical treatments for melasma. Participants will be randomly assigned to receive either triple combination cream (hydroquinone 2% + tretinoin 0.025% + fluocinolone acetonide 0.01%) or 30% metformin gel, applied once nightly for 12 weeks. All participants will use broad-spectrum sunscreen (SPF ≥30) during the daytime throughout the treatment period. Melasma severity will be assessed using the Melasma Area and Severity Index (MASI), and the study will determine which treatment is more effective and better tolerated at the end of 12 weeks.

DETAILED DESCRIPTION:
This randomized, parallel-group clinical trial will be conducted at the Department of Dermatology, Jinnah Postgraduate Medical Centre (JPMC), Karachi, Pakistan, after approval from the Institutional Review Board/Ethics Committee of JPMC. Eligible patients presenting with clinically diagnosed melasma will be screened and enrolled after obtaining written informed consent.

Participants will be randomly assigned in a 1:1 ratio to one of two treatment arms using a computer-generated randomization sequence. Group A (active comparator) will receive topical triple combination cream containing hydroquinone 2%, tretinoin 0.025%, and fluocinolone acetonide 0.01%, applied once nightly to affected facial areas for 12 weeks. Group B (experimental) will receive topical metformin gel 30%, applied once nightly to melasma-affected areas for 12 weeks. All participants in both arms will be advised to apply broad-spectrum sunscreen (SPF ≥30) during daytime throughout the treatment period.

Melasma severity will be assessed using the Melasma Area and Severity Index (MASI) at baseline and during follow-up visits over the 12-week treatment period. The primary outcome will be the proportion of participants achieving at least a 50% reduction in total MASI score from baseline at week 12. Safety and tolerability will be monitored throughout the study by documenting adverse effects reported by participants or observed on clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18- 60 years of either gender.
* Diagnosed with melasma based on clinical examination and Wood's lamp assessment.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with a history of hypersensitivity to any study medication components.
* Patients currently on other melasma treatments or those with other dermatologic conditions affecting pigmentation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with ≥50% reduction in MASI score from baseline at 12 weeks. | 12 weeks (end of treatment)
  The Melasma Area and Severity Index (MASI) will be used to assess the severity of melasma. The MASI score is calculated based on the area of involvement, darkness, and homogeneity on four facial regions. Participants achieving ≥50% reduction in total MASI score from baseline at week 12 will be classified as treatment responders. Data will be reported as the number and percentage of responders in each treatment arm and compared between arms.

SECONDARY OUTCOMES:
Mean change in MASI score from baseline to 12 weeks. | 2 weeks (end of treatment)
  MASI score will be measured at baseline and at week 12. The mean change in MASI score from baseline to week 12 will be calculated for each treatment arm.
Frequency of treatment-related adverse effects during the 12-week treatment period. | 12 weeks (during treatment)
  Adverse effects (e.g., erythema, burning, irritation, dryness) will be assessed and recorded at follow-up visits during the treatment period. Results will be summarized as the number and percentage of participants experiencing any adverse effect in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- JPMC, Karachi, Sindh, Pakistan

REFERENCES:
- [Result] Grimes PE, Pandya AG, Taylor SC, Rendon MI. Challenges in melasma treatment: need for standardization and multicenter RCTs. Dermatol Ther. 2022;35(1):e15234. doi:10.1111/dth.15234
- [Result] Steiner D, Pandya AG. Melasma and hormonal imbalance: an evidence-based review. J Eur Acad Dermatol Venereol. 2021;35(8):1630-40. doi:10.1111/jdv.17123
- [Result] Del Rosario E, Florell SR, Zone JJ. Gender and hormonal differences in melasma pathogenesis. Int J Womens Dermatol. 2023;9(2):95-103. doi:10.1016/j.ijwd.2023.02.004
- [Result] Coondoo A, Phiske M, Verma S, Lahiri K. Side-effects of topical steroids: A long overdue revisit. Indian Dermatol Online J. 2014 Oct;5(4):416-25. doi: 10.4103/2229-5178.142483. PMID 25396122
- [Result] Misitzis D, Georgala S, Katoulis AC. Comparison of the effectiveness and safety of triple combination cream vs hydroquinone monotherapy in melasma. J Cosmet Dermatol. 2022;21(9):3882-7. doi:10.1111/jocd.14278
- [Result] Frances L, Cuesta L, Leiva-Salinas M, Banuls J. Secondary mucinous carcinoma of the skin. Dermatol Online J. 2014 Apr 16;20(4):22361. PMID 24746304
- [Result] Lima EVA, Lima MA, Paixão MP, Miot HA. Assessment of the efficacy of a triple combination cream for melasma in different populations: a literature review. Clin Cosmet Investig Dermatol. 2020;13:505-10. doi:10.2147/CCID.S238536
- [Result] Pomeranz MK, Belsito DV. Mechanisms of postinflammatory hyperpigmentation and therapeutic strategies. Clin Dermatol. 2020;38(1):64-72. doi:10.1016/j.clindermatol.2019.06.009
- [Result] Lee AY. Anti-melanogenic effects of metformin: beyond diabetes. J Dermatol Sci. 2021;104(1):1-8. doi:10.1016/j.jdermsci.2021.06.002
- [Result] González-Pedraza A, Salazar-Aranda R, Pérez-Herrera P, Torres-Torres Y. Metformin as an adjuvant in dermatology: molecular mechanisms and clinical applications. Int J Dermatol. 2023;62(2):132-40. doi:10.1111/ijd.16391
- [Result] Mahmoud MMY, Kamel AM, Galal SA. Evaluation the efficacy of microneedling with topical metformin solution compared with microneedling with topical vitamin C solution in treatment of melasma. Arch Dermatol Res. 2024 Oct 5;316(9):662. doi: 10.1007/s00403-024-03355-9. PMID 39369111
- [Result] Ali Mapar M, Namdari G. Efficacy of topical metformin 15% vs placebo in melasma: RCT over 12 weeks. J Cosmet Dermatol. 2019;18(5):1357-63. doi:10.1111/jocd.12904
- [Result] Gan C, Rodrigues M. An Update on New and Existing Treatments for the Management of Melasma. Am J Clin Dermatol. 2024 Sep;25(5):717-733. doi: 10.1007/s40257-024-00863-2. Epub 2024 Jun 19. PMID 38896402
- [Result] AboAlsoud ES, Eldahshan RM, AbouKhodair Mohammed H, Elsaie ML. Safety and efficacy of topical metformin 30% cream versus triple combination cream (Kligman's formula) in treating melasma: A randomized controlled study. J Cosmet Dermatol. 2022 Jun;21(6):2508-2515. doi: 10.1111/jocd.14953. Epub 2022 Apr 9. PMID 35357753
- [Result] Mapar MA, Hemmati AA, Namdari G. Comparing the efficacy of topical metformin and placebo in the treatment of melasma: a randomized, double-blind clinical trial. J Pharm Res Int. 2019;30(4):1-8. doi:10.9734/JPRI/2019/v30i430276
- [Result] Banavase Channakeshavaiah R, Andanooru Chandrappa NK. Topical metformin in the treatment of melasma: A preliminary clinical trial. J Cosmet Dermatol. 2020 May;19(5):1161-1164. doi: 10.1111/jocd.13145. Epub 2019 Sep 10. PMID 31502392
- [Result] Mongkhon P, Ruengorn C, Awiphan R, Phosuya C, Ruanta Y, Thavorn K, Jamjanya S, Chuamanochan M, Nochaiwong S. Efficacy and safety of metformin for melasma treatment: a systematic review and meta-analysis. Front Pharmacol. 2023 Dec 13;14:1281050. doi: 10.3389/fphar.2023.1281050. eCollection 2023. PMID 38192412
- [Result] Ahmad Nasrollahi S, Sabet Nematzadeh M, Samadi A, Ayatollahi A, Yadangi S, Abels C, Firooz A. Evaluation of the safety and efficacy of a triple combination cream (hydroquinone, tretinoin, and fluocinolone) for treatment of melasma in Middle Eastern skin. Clin Cosmet Investig Dermatol. 2019 Jun 10;12:437-444. doi: 10.2147/CCID.S202285. eCollection 2019. PMID 31354327
- [Result] Atwa MA, Ahmed AH, Nada HA, Refaey SM, Jafferany M, Elsaie ML. Combined chemical peels versus trichloroacetic acid (TCA) for treating melasma: a split face study. J Dermatolog Treat. 2022 Mar;33(2):959-964. doi: 10.1080/09546634.2020.1793888. PMID 32649234
- [Result] Passeron T. Melasma pathogenesis and updated treatment options. J Eur Acad Dermatol Venereol. 2022;36(6):859-68. doi:10.1111/jdv.18101
- [Result] Neagu N, Conforti C, Agozzino M, Marangi GF, Morariu SH, Pellacani G, Persichetti P, Piccolo D, Segreto F, Zalaudek I, Dianzani C. Melasma treatment: a systematic review. J Dermatolog Treat. 2022 Jun;33(4):1816-1837. doi: 10.1080/09546634.2021.1914313. Epub 2022 Mar 23. PMID 33849384
- [Result] Rahman A, Basit A, Mohsin S, Ahmed N, Tahir M, Ishfaq A. Quality of life of melasma patients in Pakistan. Pak Armed Forces Med J. 2022;72(1):307-10.
- [Result] Handel AC, Miot LD, Miot HA. Melasma: a clinical and epidemiological review. An Bras Dermatol. 2014 Sep-Oct;89(5):771-82. doi: 10.1590/abd1806-4841.20143063. PMID 25184917
- [Result] Kang HY, Ortonne JP. Melasma update. Acta Dermatovenerol Alp Pannonica Adriat. 2009;18(2):137-42